CLINICAL TRIAL: NCT04626648
Title: Intraoperative Pauses in Relation to Stress Assessment Among Surgeons
Acronym: SAFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Eva Angenete, Professor, Sahlgrenska University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SAFT
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Stress

STUDY DESIGN:
Intervention Model Description: A randomized controlled cross-over trial was conducted in a simulator environment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery without intraoperative pause (No Intervention): Surgical procedure without pause
- Surgery with intraoperative pause (Experimental): Three-minute long intraoperative pause, including a sugar-containing drink
  Interventions: Behavioral: Pause with a sugar containing drink

INTERVENTIONS:
Behavioral: Pause with a sugar containing drink — Three-minute long intraoperative pause, including a sugar-containing drink
  Arms: Surgery with intraoperative pause

SUMMARY:
Intraoperative stress among the surgical team can be a threat to patient safety and good teamwork. During surgery, surgeons often work under stressful conditions. Reducing intraoperative stress for surgeons could benefit surgeons and subsequently patients. Based on the hypothesis that an intraoperative pause including a sugar-containing drink would decrease surgeon's stress levels, the aim of this study is to compare stress levels, in relation to intraoperative stress and how this is affected by a pause including a sugar-containing drink in simulated operations.

DETAILED DESCRIPTION:
A randomized controlled cross-over trial was conducted in a simulator environment. Primary endpoint was intra-individual change in salivary cortisol between simulations with or without a pause including a sugar containing drink. Secondary endpoints were change in heart rate, change in self-perceived stress measured by the State Trait Anxiety Inventory (STAI), and experience of the intraoperative pause.

ELIGIBILITY:
Inclusion Criteria:

* Surgeon within five years of specialization with basic laparoscopic skills, able to perform an appendectomy

Exclusion Criteria:

* diabetes
* Addison's disease
* medication with steroids or medication that affect heart rate (beta-blockers, calcium antagonists, antiarrhythmics, and digitalis) Smoking

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Salivary cortisol | 10 minutes
  Intra-individual change in salivary cortisol between simulations with or without a pause including a sugar containing drink.

SECONDARY OUTCOMES:
Heart rate | 3 hours
  Change in heart rate during surgery
self-perceived stress | 10 minutes
  measured by the State Trait Anxiety Inventory (STAI) Each STAI item is given a weighted score of 1 to 4. A rating of 4 indicates the presence of a high level of anxiety for ten S-Anxiety items and eleven T-Anxiety items. A high rating indicates the absence of anxiety for the remaining ten S-Anxiety items and nine T-Anxiety items.
Experience of the intraoperative pause. | 10 minutes
  Questionnaire with self-experience questions - no scale

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Surgery, Sahlgrenska University Hospital/Ostra, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Erestam S, Bock D, Andersson AE, Haglind E, Park J, Angenete E. The perceived benefit of intraoperative stress modifiers for surgeons: an experimental simulation study in volunteers. Patient Saf Surg. 2021 May 29;15(1):23. doi: 10.1186/s13037-021-00294-6. PMID 34051829